CLINICAL TRIAL: NCT06864052
Title: A Randomized, Open-label, Investigator-led, Pilot Trial Investigating the Incidence of New-brain Lesions on Brain MRI and Safety Between Edoxaban and Apixaban in Patients with Stroke and Nonvalvular Atrial Fibrillation
Brief Title: The Incidence of New-brain Lesions on Brain MRI and Safety Between Edoxaban and Apixaban in Patients with Stroke and Nonvalvular Atrial Fibrillation
Acronym: APIXABAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Tae-Jin Song, MD, PhD, Cerebrovascular hospital, the director of a hospital, Ewha Womans University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEUMC 2024-08-070
Record Dates: First submitted 2025-02-10; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: Non-Vitamin K Antagonist Oral Anticoagulants; Edoxaban; Apixaban
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of Apixaban (Experimental): The intervention group will receive Apixaban 2.5mg or Apixaban 5mg
  Interventions: Drug: Administration of Apixaban
- Administration of Edoxaban (Other): The control group will receive Edoxaban 15mg or 30mg or 60mg
  Interventions: Drug: Administration of Edoxaban

INTERVENTIONS:
Drug: Administration of Apixaban — Apixaban 2.5mg BID or Apixaban 5mg BID
  Arms: Administration of Apixaban
Drug: Administration of Edoxaban — Edoxaban 15mg QD or Edoxaban 30mg QD or Edoxaban 60mg QD
  Arms: Administration of Edoxaban

SUMMARY:
This study aims to determine whether there is a difference in brain lesion occurrence and safety when brain MRI is followed up between edoxaban and apixaban in stroke patients with nonvalvular atrial fibrillation through exploratory clinical trials.

DETAILED DESCRIPTION:
This study is a prospective open randomized clinical trial that can confirm which group the subject was assigned to.After randomization, either the test group or the control group is prescribed, and the outcome variable is checked at 24 months. Therefore, patients who were previously administering edoxaban and apixaban can participate in the study, but if a patient who is administering edoxaban is assigned to apixaban, the drug is taken as apixaban, and similarly, if a patient who is administering apixaban is assigned to an edoxaban, the drug is changed to edoxaban and taken. During clinical trials, testers and researchers carefully observe the occurrence of adverse reactions during the follow-up period after randomization, and closely observe outcome variables, including neurological changes. During the clinical trial period, visits are made after 6, 12, 18, and 24 months, respectively, to check the signs of physical vitality, drug history, side effects, and other research-related events, and brain MR is performed at the 24th month to check the effectiveness and safety. Brain MR can be performed for various reasons before 24 months.In the brain image performed 24 months ago, if the drug is changed or stopped for a long time, the tester plans to first implement appropriate medical measures and then determine whether to continue this study. This clinical trial is a prospective open study and will be conducted in compliance with the usual diagnosis and treatment process, and in particular, all subjects will be properly tested and treated in accordance with the standard treatment guidelines for ischemic stroke during the clinical trial.

Subjects may receive active treatment according to the standard treatment guidelines for ischemic stroke during the clinical trial. In stroke patients with nonvalvular atrial fibrillation, NOAC administration is itself a standard practice guideline, so participating in this study does not deviate from the standard treatment guidelines for stroke at all. In principle, when all planned visits are completed, the subject's participation in the clinical trial will be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 or over.
2. Patients who are neurologically stable 14 days after diagnosis of ischemic stroke and who have undergone brain MRI (including MR diffusion, FLAIR, and GRE sequence) at diagnosis of ischemic stroke (In general, the patient's condition stabilizes within seven days of acute cerebral infarction, but cerebral infarction with atrial fibrillation is more frequent than patients without atrial fibrillation, so we want to target patients with neurological stability after 14 days. Most NOAC-related clinical trials were conducted when the patient's condition became neurologically stable at least two weeks after the stroke.)
3. Patients with atrial fibrillation confirmed by 12-lead electrocardiogram or Holter's examination for more than 24 hours and nonvalvular atrial fibrillation
4. A person who voluntarily agrees to participate in this clinical trial in writing

Exclusion Criteria:

1. Patients unable or contraindicated to administer anticoagulants and antithrombotic agents
2. Patients with less than 80,000 platelets, less than 8.0 hemoglobin, liver levels, and total bilirubin levels three times the normal level in the laboratory
3. A person who is confirmed to be undergoing renal replacement treatment such as dialysis due to acute or terminal nephropathy during screening
4. A person who has been diagnosed with cancer within 6 months at the time of screening or has been treated for cancer has been confirmed to have recurrent or metastatic cancer.
5. A person who has been confirmed to be taking medication for liver diseases such as liver cirrhosis during screening
6. A person who is pregnant and nursing. However, women of childbearing age can participate only if it is certain that they are not pregnant. Women of childbearing age are defined as women except those who have not clearly undergone menopause or are unable to conceive by surgical procedures.
7. A patient with a history of hemorrhagic tendencies, gastrointestinal hemorrhage
8. Patients who have difficulty explaining and expressing their opinions on participation in the study due to decreased consciousness at the time of acquisition of consent
9. A person who judges that the tester is not appropriate for participation in the clinical trial for other reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain MR findings (Differences in the incidence of new brain lesions) | 24 months
  Brain MR findings evaluated at 24 months after the first dose of clinical trial-related drugs (new cerebral infarction (including asymptomatic), white matter hyperintensity, microhemorrhage, etc.)

SECONDARY OUTCOMES:
Major cardio-cerebrovascular events | 12 and 24 months
  Major cardio-cerebrovascular events that occurred within 12 and 24 months after the first dose of the clinical trial-related drug
Modified Rankin scale | 12 and 24 months
  Modified Rankin scale evaluated at 12 months and 24 months after the first dose of clinical trial-related drugs.
  Modified Rankin scale is a total of 7 points scale (0-6). 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
NIHSS (National Institute of Health Stroke Scale) | 12 and 24 months
  Changes in NIHSS evaluated at 12 and 24 months after first dose of clinical trial-related drug.
  NIHSS scale is a total of 43 points scale (0-42) This scale means that the lower the score, the better the prognosis, and the higher the score, the higher the possibility of disability.
Other finding of brain MR (Differences in the incidence of new brain lesions) | 24 months
  Other finding of brain MR performed 24 months after the first administration of the clinical trial-related drug (cerebrovascular findings, superficial siderosis, brain volume, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No